CLINICAL TRIAL: NCT04130958
Title: Circuit-Based Approach to Suicide: Biomarkers, Predictors, and Novel Therapeutics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P002288
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Episode; Borderline Personality Disorder; Suicide
Keywords: Transcranial Magnetic Stimulation; Intermittent Theta Burst
MeSH Terms: conditions — Borderline Personality Disorder; Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- MDE and Active iTBS-TMS (Experimental): This group will consist of patients diagnosed with MDE that are receiving active iTBS-TMS.
  Interventions: Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Active)
- BPD and Active iTBS-TMS (Experimental): This group will consist of patients diagnosed with BPD that are receiving active iTBS-TMS.
  Interventions: Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Active)
- MDE and Sham iTBS-TMS (Sham Comparator): This group will consist of patients diagnosed with MDE that are receiving sham iTBS-TMS.
  Interventions: Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Sham)
- BPD and Sham iTBS-TMS (Sham Comparator): This group will consist of patients diagnosed with BPD that are receiving sham iTBS-TMS.
  Interventions: Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Sham)

INTERVENTIONS:
Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Active) — iTBS-TMS is a noninvasive neuromodulation technique that uses a powerful magnet to induce focal electrical currents in target brain regions.
  Other Names: Active iTBS-TMS
  Arms: BPD and Active iTBS-TMS; MDE and Active iTBS-TMS
Device: Intermittent Theta Burst Transcranial Magnetic Stimulation (Sham) — The sham version of iTBS-TMS involves placing the magnet over the same target brain region but the device will not be turned on during the treatment. There will be two electrodes placed on the scalp that mimic the sensation of iTBS-TMS but does not induce focal electrical currents.
  Other Names: Sham iTBS-TMS
  Arms: BPD and Sham iTBS-TMS; MDE and Sham iTBS-TMS

SUMMARY:
This neuroimaging study is a clinical trial investigating the effectiveness of intermittent theta-burst transcranial magnetic stimulation (iTBS-TMS) to the inferior parietal lobule (IPL) in reducing suicide risk in patients with major depressive episode (MDE) or borderline personality disorder (BPD).

DETAILED DESCRIPTION:
This neuroimaging study aims to determine the effectiveness of iTBS-TMS to the IPL in reducing suicide risk in patients with MDE or BPD. This study also aims to identify the structural and functional circuit properties that characterized the suicidal brain and the signatures that explain the clinical severity of suicidal risk. Moreover, this study aims to determine biological and dimensional predictors of anti-suicidal response to iTBS-TMS and its mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Diagnosed with BPD or MDE
* Chief complaint of suicidal thoughts and behaviors

Exclusion Criteria:

* Neurological conditions with known structural brain lesion
* Prior neurosurgical procedure
* Metal in the body that is ferromagnetic or metal injury to the eyes
* Epilepsy
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt
* Psychopathology not appropriate for the treatment (e.g., manic episode or psychosis)
* Current alcohol dependence or active symptoms of non-alcohol psychoactive substance use withdrawal, as indicated by self-report
* Inability to meet the safety criteria for MRI scanning according to the protocols of the MGH Department of Radiology
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Functional Connectivity of Key Nodes | Through Treatment Completion, Average of 3 Days
  Measured using Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD/PhD, Principal Investigator — 6177265348
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No